CLINICAL TRIAL: NCT07178028
Title: ''The Agreement Between Face-to-face and Tele-assessment of Fullerton Advanced Balance (FAB) Scale in Older People''
Acronym: FAB
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Assoc. Prof., Istanbul University - Cerrahpasa
Other Study IDs: E-38981562-300-1300842
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-06

CONDITIONS: Fall Risk Assessment; Tele-assessment Reliability; Geriatric Population
Keywords: Fullerton Advanced Balance Scale; Telehealth; Fall risk; Tele-assessment; Older adults; Balance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older Adults ≥65 (Single Cohort): Single cohort of individuals aged 65 and older, residing in Istanbul and affiliated with institutions under the Darülaceze Presidency. Participants will undergo both face-to-face and tele-assessment in a randomized crossover design.

SUMMARY:
The purpose of this study is to examine the measurement consistency and reliability of the Fullerton Advanced Balance Scale (FAGBS) between the tele-assessment method and the face-to-face assessment method. In line with increasing telehealth applications, researching the remote applicability of balance assessment tools is clinically important. In this context, the remote applicability of the FAGBS will be evaluated based on measurement comparability and participant experience. Research Design: This study is an observational, cross-sectional, methodological research conducted using a randomized crossover design. Measurement consistency and reliability will be compared between two different application methods (tele-assessment and face-to-face) of a measurement tool.

Hypotheses:

H₀: There is no significant consistency in terms of measurement between the tele-assessment method and the face-to-face assessment method of the Fullerton Advanced Balance Scale.

H₁: There is a significant level of consistency in measurement between the tele-assessment method and the face-to-face assessment method of the Fullerton Advanced Balance Scale.

Participants will be randomly assigned to first undergo the FAGBS using either the face-to-face or tele-assessment method, and then reassessed using the other method within 7 days. All applications will be conducted by the same physical therapist; tele-assessment will be conducted simultaneously via the Zoom platform, and sessions will be recorded. Inter-measure consistency will be assessed using ICC, error levels using SEM and MDC, and inter-method measurement agreement using Bland-Altman analysis. Convergent validity will be assessed using the FES-I (Falls Efficacy Scale - International). Additionally, feasibility, test completion rate, and participant satisfaction will be evaluated using a questionnaire. Expected Contributions: This research will provide scientific evidence that FAGBS can be applied validly and reliably using a tele-assessment method. Thus, it will enable the remote assessment of fall risk in elderly individuals in situations where face-to-face access is limited. The study will provide meaningful contributions to the standardization and integration of tele-assessment applications into clinical practice in the field of physical therapy.

DETAILED DESCRIPTION:
Research Design:

This is an observational, cross-sectional methodological study examining the measurement consistency and reliability between tele-assessment and face-to-face applications of the Fullerton Advanced Balance Scale (FAGBS). The study will use a randomized crossover design, with data collection planned between September and January 2026.

Sample:

Participants will be individuals aged 65 and older living in Istanbul and affiliated with institutions under the Darülaceze Presidency. Purposive sampling will be used, and recruitment will occur through the university's physical therapy unit, hospital waiting areas, neighborhood pharmacies, municipal senior centers, and social networks. Participation is voluntary.

The sample size was calculated using an ICC-based hypothesis testing approach (Walter et al., 1998) assuming an expected ICC of 0.90, a minimum acceptable ICC of 0.75, α = 0.05, and 90% power. A minimum of 44 participants is required; accounting for 15% attrition, the target sample size is 52.

Assessment Procedures:

All assessments will be performed by the same physical therapist following a standardized protocol. Face-to-face assessments will take place at the Department of Physical Therapy and Rehabilitation at Istanbul University-Cerrahpaşa or Darülaceze institutions. Tele-assessments will be conducted synchronously via Zoom or WhatsApp. Participants will be randomized to either face-to-face assessment followed by tele-assessment, or vice versa, with a 7-day interval between repeated tele-assessments.

Participants will receive instructions on device setup, camera positioning, and safety measures. A companion is recommended for safety, and sessions may be video recorded with consent. Assessments will be conducted in a quiet, well-lit area with a non-slip floor, and the camera positioned approximately 2-3 meters away to capture full-body movements. Participants without compatible devices will be provided with a computer and technical guidance. Assessments will be paused if fatigue, dizziness, or fall risk occurs. Physical performance tests are brief (~10 minutes), and a rest period of 1.5-2 hours will be scheduled between assessments, extendable if needed. Internet interruptions will be managed with reconnection attempts and rescheduling if necessary.

Statistical Analysis:

Data will be analyzed using SPSS 24.0. Reliability between tele-assessment and face-to-face FAGBS applications will be evaluated using the Intraclass Correlation Coefficient (ICC), including inter-observer reliability for tele-assessment. Measurement consistency will be assessed via Bland-Altman analysis. Standard Error of Measurement (SEM) and Minimal Detectable Change (MDC) will be calculated for measurement sensitivity. Concurrent validity between FAGBS and FES-I scores will be examined using Spearman's correlation. Participant satisfaction, completion rates, and Telehealth Usability Questionnaire results will be reported descriptively (mean, standard deviation, frequency, and percentage).

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years of age or older
* Able to walk independently, even if using an assistive device
* Having a Mini-Mental State Examination (MMSE) score of ≥ 24
* Having adequate vision and hearing (able to read and understand test instructions and information materials)
* Having the necessary technical equipment and a suitable environment to participate in video conference assessments
* Providing voluntary written informed consent

Exclusion Criteria:

* History of acute conditions in the past month that may temporarily affect balance (e.g., lower limb trauma, ankle sprain, acute vestibular problems)
* History of advanced neurological diseases such as Parkinson's disease, multiple sclerosis, or stroke sequelae
* Serious orthopedic problems limiting lower limb function (e.g., recent surgery, significant movement restriction)
* Systemic medical instability that may affect balance, such as uncontrolled diabetes or advanced heart failure
* Psychiatric disorders severe enough to significantly impair communication or the assessment process
* Insufficient technical equipment, environmental support, or social resources to participate in the tele-assessment process

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study will recruit community-dwelling older adults aged 65 years and above who are able to walk without assistance or with an assistive device. Participants must have a Mini-Mental State Examination (MMSE) score of 24 or higher and possess adequate vision and hearing to understand test instructions. They must also have access to the necessary technology and environment to participate in video-based tele-assessment. Individuals with recent acute conditions affecting balance, advanced neurological or orthopedic disorders, significant systemic medical instability, severe psychiatric illness, or insufficient technical/social support for tele-assessment will be excluded.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Fullerton Advanced Balance Scale | Baseline and 7 days after first assessment
  The Fullerton Advanced Balance Scale (FABS) is a performance-based tool that measures functional balance in older adults. It consists of 10 items scored from 0-4 points, with a total score range of 0-40. Higher scores indicate better balance. The scale assesses components such as static and dynamic balance, anticipatory and reactive postural control. Assessments will be administered by a trained physical therapist in both face-to-face and tele-assessment formats.

SECONDARY OUTCOMES:
Completion rate | During tele-assessment session (Day 1)
  The proportion of participants who fully complete the tele-assessment session will be recorded. Completion is defined as finishing all items of the Fullerton Advanced Balance Scale (FABS) without discontinuation. The rate will be reported as a percentage of enrolled participants.
Participant Satisfaction Survey | Immediately after completion of the tele-assessment
  A 5-item Likert-type survey will be used to evaluate participants' experience with the tele-assessment. Items assess clarity of instructions, physical feasibility, presence of technical difficulties, overall satisfaction, and willingness to use the method again. Each item is rated on a 5-point scale (1 = strongly disagree to 5 = strongly agree). Higher scores indicate greater satisfaction.
The Telehealth Usability Questionnaire (TUQ) | Immediately after completion of the tele-assessment
  The Telehealth Usability Questionnaire (TUQ) will assess participants' perceptions of the usability of the tele-assessment system. TUQ is a validated self-report measure with multiple domains, including clarity of the interface, technical adequacy, communication quality, user satisfaction, and overall preference. Each item is rated on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree), with higher scores indicating better usability.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Zengin Alpözgen, Assoc. Prof., Study Director — İstanbul University - Cerrahpaşa
Locations (1):
- Sağlık Bilimleri Fakültesi, Istanbul, Büyükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rose DJ, Lucchese N, Wiersma LD. Development of a multidimensional balance scale for use with functionally independent older adults. Arch Phys Med Rehabil. 2006 Nov;87(11):1478-85. doi: 10.1016/j.apmr.2006.07.263. PMID 17084123
- [Background] Klein PJ, Fiedler RC, Rose DJ. Rasch Analysis of the Fullerton Advanced Balance (FAB) Scale. Physiother Can. 2011 Winter;63(1):115-25. doi: 10.3138/ptc.2009-51. Epub 2011 Jan 20. PMID 22210989
- [Background] Jasper A, Karim R, Vitente AC, Rafael CM, Tayag E, Uy SJM, Baloy RK, Lazaro R. Concurrent Validity and Reliability of In-Person and Supervised Remote STEADI Fall Risk Assessment in Community-Dwelling Older Adults. J Geriatr Phys Ther. 2025 Jan 27. doi: 10.1519/JPT.0000000000000446. Online ahead of print. PMID 39868692
- [Background] Chan JKY, Klainin-Yobas P, Chi Y, Gan JKE, Chow G, Wu XV. The effectiveness of e-interventions on fall, neuromuscular functions and quality of life in community-dwelling older adults: A systematic review and meta-analysis. Int J Nurs Stud. 2021 Jan;113:103784. doi: 10.1016/j.ijnurstu.2020.103784. Epub 2020 Oct 3. PMID 33120138